CLINICAL TRIAL: NCT04018222
Title: Translation of a Diagnostic Test for Lupus Flare Prediction From Bench to Clinic
Acronym: TOTAL FEEDBACK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progentec Diagnostics, Inc. (Industry)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: OCAST-OARS AR18-019
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: System; Lupus Erythematosus; Lupus Erythematosus; SLE; Lupus Flare
Keywords: Systemic Lupus Erythematosus; SLE; Lupus Flare; Flare Prediction; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will submit blood samples beyond what is required for standard of care treatment of Systemic Lupus Erythematosus. The additional blood samples (6 tubes, approximately 9 or 10 teaspoons of blood) will be used for blood-protein evaluation and DNA extraction.
  Blood samples are the only biospecimens that will be collected for this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lupus Cases: This cohort of patients will involve individuals with a confirmed medical history of Systemic Lupus Erythematosus. Qualified individuals will satisfy all Inclusion/Exclusion criteria.
- Healthy Controls: This cohort of patients will involve individuals whom do not have a diagnosis of Systemic Lupus Erythematosus or any other rheumatological or auto-immune diseases. Qualified individuals will satisfy all Inclusion/Exclusion criteria.

SUMMARY:
This study is investigating the development of a diagnostic test intended to predict flares in patients with Systemic Lupus Erythematosus. Over a six-month period, the participant will donate blood samples for researchers to evaluate the types of proteins that are in their blood. During this time the participant will also visit a research physician to undergo a physical exam that will include an evaluation of the disease's level of activity. Questionnaires will be answered too, either via email, phone call, or a research app for android and iPhone devices. During this six-month period, if the participant experiences a lupus flare, they are strongly encouraged to visit the research physician to receive a complimentary medical evaluation.

DETAILED DESCRIPTION:
The purpose of this study is to further validate an algorithm used in a lupus flare-prediction that has been developed. The investigators will be looking at different proteins in the blood that are commonly associated with lupus flares and could warn of the risk of a future flare. Participation in this study will involve three separate visits with a research physician for six months. These will proceed as a baseline visit, a three-month visit, and a six-month visit. During each of these visits the physician assesses the participant's physical condition and take blood samples for both research and medical purposes. Throughout this study, the participant will also complete a series of questionnaires to assess their wellness and day-to-day challenges. After the initial visit, the participant will be contacted to complete a monthly survey that evaluates if there have been any changes in your condition. This survey can be completed either via email, a phone call discussion, or the study's unique research app. Three of these six surveys will be completed during the physician's visit, however, the other three will be completed in the preferred medium. Throughout the six-month period while you are on this study, if at any point the participant experiences a flare, they are encouraged to visit the research physician. During this visit, they will receive a physician's evaluation to ensure your medical condition and collect blood samples for our research at no cost to the participant.

ELIGIBILITY:
INCLUSION CRITERIA:

Lupus Patients

* Females or males age 18 or older
* Meet ≥ 4 American College of Rheumatology (ACR) classification criteria for SLE, by medical record review and/or clinical/laboratory assessment OR
* Meet ≥ 4 Systemic Lupus Collaborating Clinic (SLICC) classification for SLE, including at least one clinical and one immunologic criterion, by medical record review and/or clinical/laboratory assessment OR
* Meet SLE classification by SLICC with ANA positivity
* Have a clinical diagnosis of active SLE, per physician assessment
* Have the ability to understand the requirements of the study, provide written informed consent including consent for the use and disclosure of research-related health information, and comply with the study data collection procedures

Healthy Controls

* Matched to a currently-enrolled patient that is self-reported race, gender, and current age within 5 years.
* No medical history of rheumatological or auto-immune diseases.

EXCLUSION CRITERIA:

* Active diagnosis of Lupus Nephritis
* Inability to comply with the study data collection procedures
* Currently being treated with cyclophosphamide
* Treated with rituximab within the last six months
* Currently being treated with an investigational drug
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with Systemic Lupus Erythematosus will comprise the study population. These patients will satisfy all inclusion/exclusion criteria for study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
SLEDAI | Baseline Physician Visit
  Systemic Lupus Erythematosus Disease Activity Index - measures the patient's disease activity through clinical and laboratory values
SLEDAI | Three-month Physician Visit
  Systemic Lupus Erythematosus Disease Activity Index - measures the patient's disease activity through clinical and laboratory values
SLEDAI | Six-month Physician Visit
  Systemic Lupus Erythematosus Disease Activity Index - measures the patient's disease activity through clinical and laboratory values

SECONDARY OUTCOMES:
SF-36 | Baseline at Physician Visit
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month One via Preferred Medium
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month Two via Preferred Medium
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month Three at Physician Visit
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month Four via Preferred Medium
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month Five via Preferred Medium
  Short Form 36 Questions. General Wellness measurement
SF-36 | Month Six at Physician Visit
  Short Form 36 Questions. General Wellness measurement

CONTACTS AND LOCATIONS:
Overall Officials: Eldon Jupe, Ph.D., Principal Investigator — Progentec Diagnostics, Inc.
Locations (3):
- United States (3):
  - IRIS Research and Development, Fort Lauderdale, Florida
  - Arthritis and Pain Associates of PG County, Greenbelt, Maryland
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munroe ME, Vista ES, Guthridge JM, Thompson LF, Merrill JT, James JA. Proinflammatory adaptive cytokine and shed tumor necrosis factor receptor levels are elevated preceding systemic lupus erythematosus disease flare. Arthritis Rheumatol. 2014 Jul;66(7):1888-99. doi: 10.1002/art.38573. PMID 24578190
- [Background] Munroe ME, Vista ES, Merrill JT, Guthridge JM, Roberts VC, James JA. Pathways of impending disease flare in African-American systemic lupus erythematosus patients. J Autoimmun. 2017 Mar;78:70-78. doi: 10.1016/j.jaut.2016.12.005. Epub 2017 Feb 2. PMID 28162788
- See also: Link to Progentec's website — https://www.progentec.com/